CLINICAL TRIAL: NCT02240849
Title: Effectiveness of Functionally Customized Pillow on Neck Pain, Disability, Quality of Sleep and Life: Randomized Controlled Trial
Brief Title: Effectiveness of Functional Pillow on Neck Pain, Disability, Quality of Sleep and Life
Acronym: EPNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, Dr, Jaseng Hospital of Korean Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JS-CT-2014-03
Record Dates: First submitted 2014-08-28; First posted 2014-09-16 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Neck Pain; Posterior Cervical Pain; Sleep Disorders
Keywords: Neck pain; functional pillow; sleep; cervical lordosis
MeSH Terms: conditions — Neck Pain; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional pillow (Experimental): cervical pillow, designed functionally to decrease neck pain and help to ensure the right support of the cervical curve, was applied to patients' posterior neck area.
  Interventions: Device: Functional pillow
- General pillow (Placebo Comparator): Applicants Randomly allocated to this group were issued by placebo-general pillow. There is not any specific intervention for their neck discomfort except for that.
  Interventions: Device: Placebo general pillow

INTERVENTIONS:
Device: Functional pillow — streamlined shape for cervical lordosis memory foam pillow functional design considered several sleep position
  Other Names: Functional pillow (Jaseng-chuna pillow™)
  Arms: Functional pillow
Device: Placebo general pillow
  Arms: General pillow

SUMMARY:
The purpose of this study is to investigate the effects of functional cervical pillow on inpatients with neck discomfort.

DETAILED DESCRIPTION:
50 inpatients with neck discomfort(NRS>4) will be randomly allocated to 2 groups. The experimental group was treated with functional cervical pillow and the control group was treated with general pillow. All applications of pillow were limited to 3-4 weeks. Primary outcomes were measured using the VAS scale. Post-treatment follow-up will be performed to measure primary outcomes at baseline, 3 day, per weeks until the duration of admission. Satisfaction levels of the patient's current status, Neck disability Index(NDI) PSQI, EQ-5D will also be collected. The applicants will also get thru the diagnosis of range of motion by X-ray(flexion, neutral, extension of their neck position)

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a Korean Medicine hospital
* Age between 18 and 69
* NRS score of >4 on the day of the intervention
* Voluntary participation with written consent given to study consent form, including cervical x-ray

Exclusion Criteria:

* Diagnosis of serious disease(s) which are possible causes of neck pain such as malignancy, vertebral fracture, spinal infection, inflammatory spondylitis, cauda-equina compression, etc.
* Prior diagnosis of other chronic disease(s) which could affect effectiveness or interpretation of treatment results such as cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, Alzheimer's disease, epilepsy, etc.
* Progressive neurologic deficit(s) or concurrent severe neurological symptoms
* Previously using any kind of functional pillow

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Neck discomfort on Visual Analogue Scale(VAS) | At baseline, 3 day, week 1, 2, 3, 4 following intervention
  The patient is asked to mark on the visual analogue scale the intensity of the neck discomfort they are experiencing during night and morning

SECONDARY OUTCOMES:
Change from baseline in Satisfaction levels on present status of him/her | At baseline, 3 day, week 1, 2, 3, 4 following intervention
  5-point Likert scale
Change from baseline in functional impairment on Neck Disability Index(NDI) | At baseline, week 2, 4 following intervention
  The NDI is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
Change from baseline in quality of sleep on Pittsburgh Sleep Quality Index(PSQI) | At baseline, week 2, 4 following intervention
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration,habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month.
Change from baseline in quality of life on EuroQol Group-5 dimension(EQ-5D) | At baseline, week 4 following intervention
  This is for checking the patients' changes on Quality of Life after using the cervical pillow
Change from baseline in radiological angle on Range of motion(ROM) | At baseline, week 4
  ROM of applicants will be assessed by X-ray diagnosis. (neutral, flexion, extension view)

CONTACTS AND LOCATIONS:
Overall Officials: Joonshik Shin, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea